CLINICAL TRIAL: NCT02909868
Title: Clinical Evaluation of Safety and Effectiveness of the BackBeat Medical Moderato System in Patients With Hypertension: A Double-Blind Randomized Trial - PV Loops Sub-study
Brief Title: CS-03 Pressure-Volume Loop Sub-study With RV Lead Positioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BackBeat Medical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CS-03 PV Loop substudy
Record Dates: First submitted 2016-09-13; First posted 2016-09-21 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RV location (Experimental): All included subjects will undergo the PV loop test with 'BackBeat PHC' ON and OFF
  Interventions: Device: BackBeat-PHC

INTERVENTIONS:
Device: BackBeat-PHC — A conductance catheter will be used to obtain PV loops prior to a Moderato pacemaker implant procedure.

SUMMARY:
The position of the RV lead may have an important role in the effectiveness of the Programmable Hypertension Control (PHC) therapy by the Moderato pacemaker eliciting a lag from which RV signals (QRS) are identified.

The study attempts to measure RV Pressure and RV Volume with PHC in two RV lead locations.

DETAILED DESCRIPTION:
Subjects found eligible for participation in the CS-03 study, who are indicated for a de novo pulse generator implant at the center participating in this sub-study and who are not 100% dependent on RV pacing are eligible for participation in this sub-study.

Patients receiving a pacemaker pulse generator exchange or who are 100% pacemaker dependent may not participate.

Eligible patients will be provided with an Informed Consent specific to this sub-study and if patients choose to participate, patients will be asked to sign the Informed Consent and will then undergo the procedures described below.

Patients will be prepared and draped for the Moderato implant procedure as detailed in the main CS-03 study protocol.

Subjects will be instrumented prior to the Moderato Pacemaker implant procedure.

The position of the RV lead will be tested at two sites known to elicit shortest QRS duration (The RV apical septum and the His region).

A series of three test periods with the Moderato System programmed to deliver predetermined PHC settings will follow.

Following the completion of these measurements, the conductance catheter will be withdrawn and the Moderato System implant will resume as described in the CS-03 protocol.

ELIGIBILITY:
Inclusion Criteria:

* Subject was included in the CS-03 study
* Subject indicated for a de novo pulse generator implant

Exclusion Criteria:

* Subject was excluded from the CS-03 study
* Subject is not 100% dependent on RV pacing
* Subject receiving a pacemaker pulse generator exchange
* Subject is unwilling or cannot provide Informed Consent for this sub study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-09-15 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in the LV volumes (ml) | up to 2 hr
  LV volume will be assessed in two RV electrode lead locations with BackBeat PHC ON and OFF
Change in the LV pressures (mmHg) | up to 2 hr
  LV pressure will be assessed in two RV electrode lead locations with BackBeat PHC ON and OFF

SECONDARY OUTCOMES:
Change in the pressure-volume ratio | up to 2 hr
  LV pressure will be assessed in two RV electrode lead locations with BackBeat PHC ON and OFF

CONTACTS AND LOCATIONS:
Overall Officials: Petr Neuzil, Prof., Principal Investigator — Na Homolce Hospital
Locations (1):
- Na Homolce Hospital, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chen CH, Fetics B, Nevo E, Rochitte CE, Chiou KR, Ding PA, Kawaguchi M, Kass DA. Noninvasive single-beat determination of left ventricular end-systolic elastance in humans. J Am Coll Cardiol. 2001 Dec;38(7):2028-34. doi: 10.1016/s0735-1097(01)01651-5. PMID 11738311
- [Background] Klotz S, Dickstein ML, Burkhoff D. A computational method of prediction of the end-diastolic pressure-volume relationship by single beat. Nat Protoc. 2007;2(9):2152-8. doi: 10.1038/nprot.2007.270. PMID 17853871